CLINICAL TRIAL: NCT03149731
Title: Monitoring of Cerebral and Abdominal Tissue Oxygen Saturation in Neonates
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Tian Li-1, Department of Anesthesiology and Perioperative Medicine, Xijing Hospital
Other Study IDs: XijingHosp
Record Dates: First submitted 2017-05-08; First posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Establish the Incidence Rate of Abdominal and Cerebral Hyperoxemia and Hypoxemia Events in Neonates at Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: NIRS — The recent technological advancement of tissue NIRS enables continuous, real time and bedside monitoring of hemoglobin oxygen saturation in mixed arterial, venous, and primarily capillary blood in the tissue bed being probed.

SUMMARY:
Near-infrared spectroscopy (NIRS) functions in a manner similar to pulse oximetry, using the difference in absorptive qualities of oxy- and deoxyhemoglobin to infrared light to quantify the percent saturation. There is also available evidence shows that tissue oximetry is sensitive and has a quicker response to physiological derangement, such as bradycardia, in preterm newborns. Additionally, it is demonstrated that reduced postoperative cerebral tissue oxygenation index variability in neonatal survivors of congenital heart disease surgery with poor neurodevelopmental outcomes. The SafeBoosC phase II randomized clinical trial hypothesizes that the burden of hypo- and hyperoxia can be reduced, and consequently the risk of brain injury, by the combined use of close monitoring of the cerebral rStO2 and an evidence-based treatment guideline to correct deviations in rStO2 outside a predefined target range. In this study, we will monitor 2 different tissue beds including cerebral and abdominal somatic tissue rStO2 and SpO2 in neonates. Further research is needed to investigate clinical implications for using this measure to drive therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Term infants (37-42 weeks of gestation)
2. Elective cesarean section after pregnancy

Exclusion Criteria:

1. Thick hair that makes good measurements difficult/impossible
2. Obvious malformations or syndrome
3. Complications in relation to the cesarean section

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 120 ASA class I or II parturients between 37 to 42 weeks of gestation with singleton vertex pregnancy and scheduled for elective cesarean delivery under spinal anesthesia.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-11-01 (Estimated); Study Completion 2018-02-01 (Estimated)

PRIMARY OUTCOMES:
Cerebral and abdominal NIRS in neonates | After birth in 20 min
  Cerebral and abdominal tissue oxygen saturation was obtained using 4-wavelength (690, 780, 805 and 850nm) near-infrared spectroscopy (FORE-SIGHT, CAS Medical Systems, Branford, CT) with a transducer containing a fiber optic emitter and one detector located 25mm from the light source. A non-adhesive optode (FORE-SIGHT sensor kit small, CAS Medical Systems, Branford, CT) was placed on the left forehead and abdomen.

SECONDARY OUTCOMES:
Pulse oximetry in neonates | After birth in 20 min
  Pulse oximetry data (SpO2) were collected in a time-synchronized fashion with the NIRS data using the transport monitor (Philips IntelliVue MMS X2 equipped with multi-measurement module, Philips Healthcare, Andover, MA) and a non-adhesive probe placed on the hand or foot (Neonatal-Adult SpO2 Sensor, Philips Healthcare, Andover, MA).

CONTACTS AND LOCATIONS:
Overall Officials: Li Tian, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Result] SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network; Carlo WA, Finer NN, Walsh MC, Rich W, Gantz MG, Laptook AR, Yoder BA, Faix RG, Das A, Poole WK, Schibler K, Newman NS, Ambalavanan N, Frantz ID 3rd, Piazza AJ, Sanchez PJ, Morris BH, Laroia N, Phelps DL, Poindexter BB, Cotten CM, Van Meurs KP, Duara S, Narendran V, Sood BG, O'Shea TM, Bell EF, Ehrenkranz RA, Watterberg KL, Higgins RD. Target ranges of oxygen saturation in extremely preterm infants. N Engl J Med. 2010 May 27;362(21):1959-69. doi: 10.1056/NEJMoa0911781. Epub 2010 May 16. PMID 20472937
- [Result] BOOST II United Kingdom Collaborative Group; BOOST II Australia Collaborative Group; BOOST II New Zealand Collaborative Group; Stenson BJ, Tarnow-Mordi WO, Darlow BA, Simes J, Juszczak E, Askie L, Battin M, Bowler U, Broadbent R, Cairns P, Davis PG, Deshpande S, Donoghoe M, Doyle L, Fleck BW, Ghadge A, Hague W, Halliday HL, Hewson M, King A, Kirby A, Marlow N, Meyer M, Morley C, Simmer K, Tin W, Wardle SP, Brocklehurst P. Oxygen saturation and outcomes in preterm infants. N Engl J Med. 2013 May 30;368(22):2094-104. doi: 10.1056/NEJMoa1302298. Epub 2013 May 5. PMID 23642047
- [Result] Spaeder MC, Klugman D, Skurow-Todd K, Glass P, Jonas RA, Donofrio MT. Perioperative Near-Infrared Spectroscopy Monitoring in Neonates With Congenital Heart Disease: Relationship of Cerebral Tissue Oxygenation Index Variability With Neurodevelopmental Outcome. Pediatr Crit Care Med. 2017 Mar;18(3):213-218. doi: 10.1097/PCC.0000000000001056. PMID 28067688
- [Result] Schmid MB, Hopfner RJ, Lenhof S, Hummler HD, Fuchs H. Cerebral oxygenation during intermittent hypoxemia and bradycardia in preterm infants. Neonatology. 2015;107(2):137-46. doi: 10.1159/000368294. Epub 2014 Dec 20. PMID 25531368